CLINICAL TRIAL: NCT03877107
Title: Effect of Depletive Lumbar Puncture and Cerebrospinal Fluid Shunt Surgery on Lower Urinary Tract Dysfunction in Normal Pressure Hydrocephalus
Brief Title: Effect of Depletive Lumbar Puncture on Lower Urinary Tract Dysfunction in iNPH
Acronym: PLHPN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: EssaiClinique_PL-HPN (Other)
Responsible Party: Sponsor-Investigator, EssaiClinique_PL-HPN, Clinical Professor, University Hospital, Grenoble
Organization: University Hospital, Grenoble (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PL HPN
Record Dates: First submitted 2019-03-13; First posted 2019-03-15 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Normal Pressure Hydrocephalus
Keywords: lower urinary tract dysfunction; urinary incontinence; normal pressure hydrocephalus; overactive bladder
MeSH Terms: conditions — Hydrocephalus, Normal Pressure; Urinary Incontinence; Urinary Bladder, Overactive

STUDY DESIGN:
Intervention Model Description: Evaluation of urinary symptoms before and after depletive lumbar puncture and after shunt surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single cohort (Other): Participants presenting at least 2/3 of symptom triad : gait disturbance, urinary symptoms and cognitive disturbance Ventricular enlargement non explained by cortical atrophy Cognitive capacity to understand the study and give informed consent (mini mental state > 13), speaking and reading french.
  Interventions: Diagnostic Test: Urinary symptoms profile questionnaire; Diagnostic Test: Micturition calendar

INTERVENTIONS:
Diagnostic Test: Urinary symptoms profile questionnaire — Validated questionnaire (international) with validated french translation, before and after lumbar puncture, and after surgery if surgery is realized
Diagnostic Test: Micturition calendar — Micturition calendar on 2 consecutive days, before and after lumbar puncture, and after surgery if surgery is realized

SUMMARY:
Lower urinary tract dysfunction in normal pressure hydrocephalus has received little attention from the scientific community. Urinary symptoms in normal pressure hydrocephalus are mainly represented by overactive bladder, which is a significant burden for the concerned patients. A harmonization of neuro-urological practices in the pre-therapeutic evaluation of patients suffering from normal pressure hydrocephalus is necessary.

The investigators conducted a bicentric prospective study aiming to evaluate the effect of depletive lumbar puncture on urinary symptoms in iNPH.

The secondary objective was to evaluate, in the same participants previously diagnosed, the effect of cerebrospinal fluid shunt surgery on urinary symptoms.

DETAILED DESCRIPTION:
Prospective study interventional but non invasive Bicentric in two universitarian hospitals in France On a cohort of patients presenting at least two out of three symptoms of the classic triad (urinary symptoms, cognitive symptoms and gait disturbance) and enlargement of ventricles non explained by cortical atrophy.

Participants are offered, as routine care, a diagnostic evaluation of the effect of depletive lumbar puncture on these triad symptoms (this exam is part of routine care).

Before the planned lumbar puncture, the participants are requested to participate to the study, with written consent and information given. The participants are requested to fill in a USP (urinary symptoms profile, validated international questionnaire) questionnaire and a micturition calendar. The same urinary evaluation is made 5 days after lumbar puncture. Gait and cognition are evaluated as in routine practice.

Of the participants initially evaluated, some will be proposed shunt surgery (routine care). These participants will be proposed to fill in the same questionnaire and micturition calendar around 3 months after shunt surgery (post operative evaluation).

ELIGIBILITY:
Inclusion Criteria:

* 2/3 symptoms triad : gait disturbance + cognitive disturbance + urinary symptoms
* Ventricular enlargement non explained by cortical atrophy

Exclusion Criteria:

* analphabetism or not french speaking
* Cognitive disability making understanding of study impossible (as informed consent)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-03-13 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Effect of depletive lumbar puncture on overactive bladder symptoms 1 | 5 days after lumbar puncture
  evaluation on USP questionnaire, subsection HAV [0-21]
Effect of depletive lumbar puncture on overactive bladder symptoms 2 | 5 days after lumbar puncture
  evaluation on micturition calendar on 2 days [number of mictions/day]

SECONDARY OUTCOMES:
Effect of shunt surgery on overactive bladder symptoms 1 | 3 to 4 months after surgery
  evaluation on micturition calendar on 2 days [number of mictions/day]
Effect of shunt surgery on overactive bladder symptoms 2 | 3 to 4 months after surgery
  evaluation on USP questionnaire, subsection HAV [0-21]

CONTACTS AND LOCATIONS:
Overall Officials: Jean Alexandre LONG, MD PHD, Study Director — University Hospital, Grenoble
Locations (2):
- France (2):
  - University Hospital of Grenoble, Grenoble
  - University Hospital of Lyon, Lyon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mary P, Gallisa JM, Laroque S, Bedou G, Maillard A, Bousquet C, Negre C, Gaillard N, Dutray A, Fadat B, Jurici S, Olivier N, Cisse B, Sablot D. [Predictive value of postural and dynamic walking parameters after high-volume lumbar puncture in normal pressure hydrocephalus]. Rev Neurol (Paris). 2013 Apr;169(4):321-7. doi: 10.1016/j.neurol.2012.09.010. Epub 2013 Feb 12. French. PMID 23415160
- [Result] Jonas S, Brown J. Neurogenic bladder in normal pressure hydrocephalus. Urology. 1975 Jan;5(1):44-50. doi: 10.1016/0090-4295(75)90300-3. PMID 1114545
- [Result] Sakakibara R, Uchida Y, Ishii K, Kazui H, Hashimoto M, Ishikawa M, Yuasa T, Kishi M, Ogawa E, Tateno F, Uchiyama T, Yamamoto T, Yamanishi T, Terada H; SINPHONI (Study of Idiopathic Normal Pressure Hydrocephalus On Neurological Improvement). Correlation of right frontal hypoperfusion and urinary dysfunction in iNPH: a SPECT study. Neurourol Urodyn. 2012 Jan;31(1):50-5. doi: 10.1002/nau.21222. Epub 2011 Oct 28. PMID 22038765
- [Result] Sakakibara R, Kanda T, Sekido T, Uchiyama T, Awa Y, Ito T, Liu Z, Yamamoto T, Yamanishi T, Yuasa T, Shirai K, Hattori T. Mechanism of bladder dysfunction in idiopathic normal pressure hydrocephalus. Neurourol Urodyn. 2008;27(6):507-10. doi: 10.1002/nau.20547. PMID 18092331
- [Result] Sakakibara R, Uchiyama T, Kanda T, Uchida Y, Kishi M, Hattori T. [Urinary dysfunction in idiopathic normal pressure hydrocephalus]. Brain Nerve. 2008 Mar;60(3):233-9. Japanese. PMID 18402070
- [Result] Campos-Juanatey F, Gutierrez-Banos JL, Portillo-Martin JA, Zubillaga-Guerrero S. Assessment of the urodynamic diagnosis in patients with urinary incontinence associated with normal pressure hydrocephalus. Neurourol Urodyn. 2015 Jun;34(5):465-8. doi: 10.1002/nau.22600. Epub 2014 Apr 12. PMID 24729303
- [Result] Kazui H, Mori E, Ohkawa S, Okada T, Kondo T, Sakakibara R, Ueki O, Nishio Y, Ishii K, Kawaguchi T, Ishikawa M, Takeda M. Predictors of the disappearance of triad symptoms in patients with idiopathic normal pressure hydrocephalus after shunt surgery. J Neurol Sci. 2013 May 15;328(1-2):64-9. doi: 10.1016/j.jns.2013.02.020. Epub 2013 Mar 16. PMID 23510566
- [Result] Mouton Paradot G, Baledent O, Sallioux G, Lehmann P, Gondry-Jouet C, Le Gars D. [Contribution of phase-contrast MRI to the management of patients with normal pressure hydrocephalus: Can it predict response to shunting?]. Neurochirurgie. 2010 Feb;56(1):50-4. doi: 10.1016/j.neuchi.2009.12.007. Epub 2010 Jan 25. French. PMID 20097391
- [Result] Sakakibara R. Lower urinary tract dysfunction in patients with brain lesions. Handb Clin Neurol. 2015;130:269-87. doi: 10.1016/B978-0-444-63247-0.00015-8. PMID 26003249
- [Result] Griffiths D, Tadic SD. Bladder control, urgency, and urge incontinence: evidence from functional brain imaging. Neurourol Urodyn. 2008;27(6):466-74. doi: 10.1002/nau.20549. PMID 18092336
- [Result] Sakakibara R, Panicker J, Fowler CJ, Tateno F, Kishi M, Tsuyusaki Y, Yamanishi T, Uchiyama T, Yamamoto T, Yano M. Is overactive bladder a brain disease? The pathophysiological role of cerebral white matter in the elderly. Int J Urol. 2014 Jan;21(1):33-8. doi: 10.1111/iju.12288. Epub 2013 Sep 30. PMID 24118122
- [Result] Sakakibara R, Uchida Y, Ishii K, Hashimoto M, Ishikawa M, Kazui H, Yamamoto T, Uchiyama T, Tateno F, Kishi M, Tsuyusaki Y, Aiba Y, Tateno H, Nagao T, Terada H, Inaoka T; Members of SINPHONI (Study of Idiopathic Normal Pressure Hydrocephalus On Neurological Improvement). Bladder recovery relates with increased mid-cingulate perfusion after shunt surgery in idiopathic normal-pressure hydrocephalus: a single-photon emission tomography study. Int Urol Nephrol. 2016 Feb;48(2):169-74. doi: 10.1007/s11255-015-1162-2. Epub 2015 Nov 17. PMID 26578001
- [Result] Kang K, Hwang SK, Lee HW. Shunt-responsive idiopathic normal pressure hydrocephalus patient with delayed improvement after tap test. J Korean Neurosurg Soc. 2013 Nov;54(5):437-40. doi: 10.3340/jkns.2013.54.5.437. Epub 2013 Nov 30. PMID 24379955
- [Result] Wikkelso C, Andersson H, Blomstrand C, Lindqvist G. The clinical effect of lumbar puncture in normal pressure hydrocephalus. J Neurol Neurosurg Psychiatry. 1982 Jan;45(1):64-9. doi: 10.1136/jnnp.45.1.64. PMID 7062072
- [Result] Lim TS, Yong SW, Moon SY. Repetitive lumbar punctures as treatment for normal pressure hydrocephalus. Eur Neurol. 2009;62(5):293-7. doi: 10.1159/000235808. Epub 2009 Aug 27. PMID 19713705
- [Result] Ahlberg J, Norlen L, Blomstrand C, Wikkelso C. Outcome of shunt operation on urinary incontinence in normal pressure hydrocephalus predicted by lumbar puncture. J Neurol Neurosurg Psychiatry. 1988 Jan;51(1):105-8. doi: 10.1136/jnnp.51.1.105. PMID 3351510
- [Result] Aruga S, Kuwana N, Shiroki Y, Takahashi S, Samejima N, Watanabe A, Seki Y, Igawa Y, Homma Y. Effect of cerebrospinal fluid shunt surgery on lower urinary tract dysfunction in idiopathic normal pressure hydrocephalus. Neurourol Urodyn. 2018 Mar;37(3):1053-1059. doi: 10.1002/nau.23399. Epub 2017 Sep 11. PMID 28892272
- [Result] Krzastek SC, Bruch WM, Robinson SP, Young HF, Klausner AP. Characterization of lower urinary tract symptoms in patients with idiopathic normal pressure hydrocephalus. Neurourol Urodyn. 2017 Apr;36(4):1167-1173. doi: 10.1002/nau.23084. Epub 2016 Aug 4. PMID 27490149